CLINICAL TRIAL: NCT04549584
Title: Neoadjuvant Chemotherapy Response in Metaplastic Carcinoma of Triple Negative Breast Cancer
Acronym: NEO-SMART
Status: Terminated | Type: Observational
Why Stopped: due to poor enrolled patients
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong-Gon Moon, Medical doctor, Clinical Professor, Seoul National University Hospital
Other Study IDs: 2004-261-112
Record Dates: First submitted 2020-07-30; First posted 2020-09-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-07

CONDITIONS: Metaplastic Breast Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — tissue obtained by core needle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metaplastic breast cancer: Histologically determined to be a metaplastic breast cancer or tested positive for vimentin/Pan CK patients decides as the metaplastic breast cancer.
  Interventions: Diagnostic Test: Vimentin/pan CK stain
- non-metaplastic breast cancer: Patients with vimentin/Pan CK negative are diagnosed with non-metaplastic breast cancer

INTERVENTIONS:
Diagnostic Test: Vimentin/pan CK stain — Vimentin/pan CK stain positive/negative
  Groups: metaplastic breast cancer

SUMMARY:
prospective study for response of neoadjuvant chemotherapy in metaplastic carcinoma of triple negative breast cancer

DETAILED DESCRIPTION:
Vimentin/Pan CK staining will be performed on tissues of patient who visited Seoul National University Hospital and were diagnosed with triple negative breast cancer and decided to perform neoadjuvant chemotherapy under clinical judgement.

Histologically determined to be a metaplastic breast cancer or tested positive for vimentin/Pan CK patients decides as the metaplastic breast cancer. They evaluate the response rate of the neoadjuvant chemotherapy.

Patients with vimentin/Pan CK negative are diagnosed with non-metaplastic breast cancer and this group also confirms the response rate of neoadjuvant chemotherapy.

The group of metaplastic breast cancer will enroll 50 people, and the group of non-metaplastic breast cancer will enroll 100 people.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* patients with triple negative breast cancer diagnosed Seoul National University Hospital
* patients who decided to perform neoadjuvant chemotherapy under clinical judgement

Exclusion Criteria:

* not applicable

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * over 20 years old
  * patients with triple negative breast cancer diagnosed Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
response rate of neoadjuvant chemotherapy | After neoadjuvant chemotherapy was finished. Average 6 month later.
  response criteria for neoadjuvant chemotherapy-complete response (CR), partial response (PR), and no response (NR)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong Gon Moon, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satelli A, Li S. Vimentin in cancer and its potential as a molecular target for cancer therapy. Cell Mol Life Sci. 2011 Sep;68(18):3033-46. doi: 10.1007/s00018-011-0735-1. Epub 2011 Jun 3. PMID 21637948
- [Background] Schwartz TL, Mogal H, Papageorgiou C, Veerapong J, Hsueh EC. Metaplastic breast cancer: histologic characteristics, prognostic factors and systemic treatment strategies. Exp Hematol Oncol. 2013 Nov 14;2(1):31. doi: 10.1186/2162-3619-2-31. PMID 24499560
- [Background] Adams S. Dramatic response of metaplastic breast cancer to chemo-immunotherapy. NPJ Breast Cancer. 2017 Mar 29;3:8. doi: 10.1038/s41523-017-0011-0. eCollection 2017. PMID 28649648